CLINICAL TRIAL: NCT04449393
Title: Effect of Enamel Matrix Derivative in the Non-surgical Treatment of Periodontal Maintenance Patients
Brief Title: Enamel Matrix Derivative in Non-surgical Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christian Wehner, DMD, Dr.med.dent., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1248/2020
Record Dates: First submitted 2020-06-20; First posted 2020-06-26 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Periodontitis
Keywords: Enamel Matrix Derivative; Periodontitis; Non-surgical periodontal therapy
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Emdogain® FL (Experimental): Non-surgical periodontal therapy in terms of scaling and root planing will be applied at sites with remaining periodontal pockets at reevaluation. EDTA gel will be applied for 2 minutes in the respective pockets, followed by rinsing with saline, drying and application of Emdogain® FL.
  Interventions: Device: Emdogain® FL
- Control group (Placebo Comparator): Non-surgical periodontal therapy in terms of scaling and root planing will be applied at sites with remaining periodontal pockets at reevaluation, followed by rinsing with saline.
  Interventions: Other: Scaling and root planing

INTERVENTIONS:
Device: Emdogain® FL — Emdogain® FL is an enamel matrix derivative intended for subgingival and topical application in conjunction with scaling and root planing procedures to provide regeneration of tooth support lost due to periodontal disease. Emdogain® FL has been shown to be effective in residual pockets with probing depths from 5mm to 9mm with no furcation involvement in patients with adequate plaque control. Emdogain® FL has also been shown to enhance the early healing of periodontal soft tissue wounds resulting from the instrumentation of periodontal pockets.
  Arms: Emdogain® FL
Other: Scaling and root planing — Scaling and root planing procedures as part of non-surgical periodontal therapy involves mechanical removal of dental plaque and calculus using curettes and sonic scalers.
  Arms: Control group

SUMMARY:
The aim of the study is to investigate the effect of enamel matrix derivative in addition to scaling and root planing in comparison to scaling and root planing only in periodontitis patients that have already undergone initial periodontal therapy and are in periodontal maintenance.

DETAILED DESCRIPTION:
Enamel matrix derivative (EMD) have already been widely applied as a regenerative bio-modulator in periodontal surgery and have been demonstrated to enhance periodontal regeneration. Recently, also its flapless, non-surgical application has been shown to have beneficial effects when applied during initial therapy of periodontitis.

The present study is designed as a single-blinded randomized controlled clinical trial. We plan to include a total of 50 periodontitis patients that have already undergone initial periodontal therapy, but still show remaining sites with increased periodontal probing depth (PPD). Patients will be randomly allocated at a 1:1 ratio to either scaling and root planing (SRP) in combination with EMD application into the affected pockets (test group, n=25) or to SRP only (control group, n=25). Before treatment, as well as after 3, 6 and 12 months, we plan to assess site-specific periodontal parameters as well as whole-mouth oral hygiene indices. Furthermore, we intend to evaluate gingival crevicular fluid, as well as parameters representing periodontal disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis stage III
* Patients that have completed initial periodontal therapy, and have remaining periodontal pockets of ≥6mm up to 9mm PPD
* Given written informed consent form for participation in the study

Exclusion Criteria:

* Systemic antibiotics within the previous 3 months
* Pregnant or breastfeeding women
* Any current or past clinically significant pathology/disease (comorbidity) that, in the opinion of the periodontists, might confound the results or poses an additional risk to the subject during participation in the study, such as renal insufficiency, malignancy, rheumatoid osteoarthritis, human immunodeficiency syndrome.
* Patients with at least one tooth of mobility grade 0 or 1 and/or furcation involvement grade 0 or I according to Hamp

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Periodontal probing depth (PPD) | At baseline
  Distance from the gingival margin to the base of the pocket with a calibrated periodontal probe
Periodontal probing depth (PPD) | After 3 months
  Distance from the gingival margin to the base of the pocket with a calibrated periodontal probe
Periodontal probing depth (PPD) | After 6 months
  Distance from the gingival margin to the base of the pocket with a calibrated periodontal probe
Periodontal probing depth (PPD) | After 12 months
  Distance from the gingival margin to the base of the pocket with a calibrated periodontal probe

SECONDARY OUTCOMES:
CAL (mm) | At baseline, after 3, 6 and 12 months
  CAL (Clinical attachment level): the probing depth and the distance from the gingival margin to the CEJ API: Approximal plaque index PBI: Papillary Bleeding Index PESA:Periodontal Epithelial Surface Area PISA: periodontal inflamed surface area GCF: Gingival crevicular fluid
API, PBI (%) | At baseline, after 3, 6 and 12 months
  API: Approximal plaque index PBI: Papillary Bleeding Index
PESA, PISA (mm2) | At baseline, after 3, 6 and 12 months
  PESA:Periodontal Epithelial Surface Area PISA: periodontal inflamed surface area
GCF markers for periodontal regeneration | At baseline, after 3, 6 and 12 months
  GCF: Gingival crevicular fluid
Periodontal bacteria | At baseline, after 3, 6 and 12 months
  Microbiologic evaluation of GCF via polymerase chain reaction (PCR) DNA probe test kit

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Dentistry Vienna, Vienna, Austria

REFERENCES:
- [Derived] Wehner C, Tur D, Durstberger G, Laky M, Laky B, Andrukhov O, Moritz A, Rausch-Fan X. Effects of enamel matrix derivative in nonsurgical periodontal therapy on pro-inflammatory profiles, microbial environment and clinical outcome: a randomized clinical trial. Clin Oral Investig. 2023 Nov;27(11):6493-6502. doi: 10.1007/s00784-023-05254-1. Epub 2023 Oct 16. PMID 37843637